CLINICAL TRIAL: NCT01294709
Title: A Double-Blind, Randomized, Placebo-Controlled, 2-Period Crossover Study to Assess the Safety, Tolerability, and Effects of MK-0974 on Exercise Tolerance in Patients With Stable Angina
Brief Title: A Study to Assess the Safety, Tolerability, and Effects of MK-0974 (Telcagepant) on Exercise Tolerance in Patients With Stable Angina (MK-0974-014)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0974-014
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Results first posted 2014-09-10 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-09

CONDITIONS: Angina Pectoris; Coronary Heart Disease; Calcitonin Gene-related Peptide Receptor
Keywords: angina pectoris; coronary artery disease; calcitonin gene-related peptide; exercise tolerance,
MeSH Terms: conditions — Angina Pectoris; Coronary Disease; Coronary Artery Disease | interventions — telcagepant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telcagepant/ Placebo (Experimental): Participants receive single oral dose of 600 mg (two 300 mg capsules or two bioequivalent 280 mg tablets) or 900 mg telcagepant (three 300 mg capsules) in Period 1 and single oral dose of two capsules or tablets of placebo for telcagepant (or three capsules of placebo for telcagepant) in Period 2 of the crossover. Each treatment period is separated by a washout of 96-240 hours.
  Interventions: Drug: telcagepant; Drug: Placebo to telcagepant
- Placebo/Telcagepant (Experimental): Participants receive single oral dose of two capsules or tablets of placebo for telcagepant (or three capsules of placebo for telcagepant) in Period 1 and a single oral dose of 600 mg (two 300 mg capsules or two bioequivalent 280 mg tablets) or 900 mg telcagepant (three 300 mg capsules) in Period 2 of the crossover. Each treatment period is separated by a washout of 96-240 hours.
  Interventions: Drug: telcagepant; Drug: Placebo to telcagepant

INTERVENTIONS:
Drug: telcagepant
  Other Names: MK-0974
Drug: Placebo to telcagepant

SUMMARY:
This study will assess the safety of telcagepant in coronary artery disease (CAD) participants with stable angina during exercise treadmill testing and evaluate whether calcitonin gene-related peptide (CGRP) receptor antagonism by telcagepant reduces exercise tolerance in these participants. Primary hypothesis is that telcagepant does not significantly decrease exercise duration compared to placebo, as measured by a treadmill exercise test; that is, the true treatment difference in exercise duration (MK-0974 - Placebo) >= -60 seconds.

DETAILED DESCRIPTION:
Amendment 3 of the protocol reduced the dose of telcagepant to be administered from a single dose of 900 mg to a single dose of 600 mg. Pooled data from both the 600-mg and the 900-mg group wiil be utilized in the analyses. Also due to supply issues regarding the 300 mg telcagepant capsules, 280 mg telcagepant tablets with demonstrated bioequivalence to the 300 mg telcagepant capsules, could be administered to participants enrolled after the implementation of Amendment 3.

ELIGIBILITY:
Inclusion:

* Participant has clinically documented stable coronary artery disease as demonstrated by coronary angiography, echocardiogram, or stress test, etc., or participant is on stable doses of current medication for the treatment of coronary artery disease for a minimum of 30 days.
* Participant has a history of stable angina (chronic stable angina pectoris that is triggered by physical effort and relieved by rest and/or sublingual nitroglycerin) for at least 3 months prior to study start, with no intervening symptoms of unstable angina.
* Participant is able to demonstrate reproducibly positive exercise tests by completing treadmill tests on 2 separate days, within 1-8 days.
* Participant agrees to refrain from drinking alcohol from 24 hours prior to study drug administration, on study procedure days, and until release from the study facility.
* Participants agrees to refrain from smoking from midnight before study procedures until study procedures are complete for the day.
* Participant has no clinically significant abnormality on screening laboratory safety assessment.
* Participant agrees to refrain from unaccustomed strenuous physical activity from the prestudy (screening) visit, throughout the study, and until the post-study visit.

Exclusion:

* Participant is pregnant (positive serum beta-human chorionic gonadotropin [β-hCG] test at prestudy), breast-feeding, or is a female expecting to conceive within the projected duration of the study. Postmenopausal women who are currently using hormone replacement therapy are excluded from participation in the study.
* Participant has electrocardiogram (ECG) findings that interfere with ECG interpretation or may cause false positive stress test (e.g., > 1 mm horizontal or downsloping ST-segment depression at rest in any standard electrocardiographic lead, Lown-Ganong-Levine syndrome, Wolff-Parkinson-White (WPW), left bundle branch block (LBBB), left ventricular hypertrophy (LVH) with repolarization abnormality, pectus excavatum, ventricular pacemaker, etc.). Note: these ECG findings may affect stress test results; there may be other findings that have not been included which may affect test results. These ECG findings are exclusions only if these findings may jeopardize interpretation of stress test results.
* Participant has heart rate-corrected QT interval (QTc) (Bazett) > 500 ms on resting ECG.
* Participant has uncontrolled high blood pressure at prestudy screening.
* Participant has a baseline heart rate of <40 or >96 beats per minute at screening.
* Participant has unstable angina, hypertrophic cardiomyopathy, valvular heart disease, congenital cardiac defect, severe aortic stenosis, class III or IV heart failure.
* Participant has diabetes and is, in the opinion of the investigator, unable to comply with the pre-and post-dosing fasting requirements of the study due to risks of hypoglycemia.
* Participant is unable to withhold acetohexamide, chlorpropamide, glimepride, glimepiride and pioglitazone, glimepride and rosiglitazone, glipizide, glipizide and metformin, glyburide, glyburide and metformin, tolazamide, tolbutamide, or any other medication, that in the opinion of the investigator is likely to result in hypoglycemia within 8 hours of dosing.
* Participant has had myocardial infarction or coronary revascularization within the prior 2 months.
* Participant has acute myocarditis or pericarditis.
* Participant is obese, with adipose tissue which may interfere with ECG interpretation, or in the opinion of the investigator, whose obesity puts the participant at medical risk.
* Participant has clinically significant hypokalemia or hypomagnesemia.
* Participant has a history of any illness that, in the opinion of the investigator, might confound the results of the study or poses an additional risk to the participant by their participation in the study.
* Participant must not have taken any of the following medications in the time frame specified: Participant is unable to refrain from or anticipates the use of any herbal remedies beginning approximately 2 weeks (or 5 half-lives) prior to administration of the initial dose of study drug, throughout the study (including washout intervals between treatments), until the post-study visit; participant is unable to refrain from taking a drug metabolized by cytochrome P450 3A4 (CYP3A4) until at least 48 hours post dose (the exact length of time a specific drug metabolized by CYP3A4 is withheld is dependent on the therapeutic index of the drug and the extent to which it is metabolized by CYP3A4); participant consumes excessive amounts of alcohol which, in the opinion of the investigator, puts the participant at medical risk by participating in the study (participant has clinical [e.g., enlarged liver] or laboratory evidence [e.g., elevated alanine aminotransferase (ALT)], of chronic alcoholism or drug abuse, in the opinion of the investigator); participants is currently a regular user (including: recreational use") of any illicit drugs or has a history of drug (including alcohol) abuse within approximately 6 months; participant has taken potent CYP3A4 inhibitors, including but not limited to cyclosporine, systemic (oral/intravenous) itraconazole, ketoconazole, erythromycin, clarithromycin, telithromycin, nefazodone, human immunodeficiency virus (HIV) protease inhibitors within 1 month prior to dosing with MK-0974 or placebo and throughout the study period; participant has taken moderate CYP3A4 inhibitors, including but not limited to verapamil, diltiazem, fluconazole, fluvoxamine, fluoxetine, aprepitant within 2 weeks prior to dosing with MK-0974 or placebo and throughout the study period; participant has taken potent CYP3A4 inducers, including but not limited to rifampicin, rifabutin, carbamazepine, phenytoin, barbiturates, systemic glucocorticoids (replacements and inhaled are permitted), nevirapine, efavirenz, pioglitazone, primidone, St. John's wort within 1 month prior to dosing MK-0974 or placebo and throughout the study period; participant has taken triptans, ergot alkaloids within 48 hours prior to dosing MK-0974 or placebo and throughout the study period; participant has taken digoxin, medications that prolong QTc interval such as Class IA and Class III anti-arrhythmics (quinidine, procainamide, amiodarone, sotalol, etc), Seldane (terfenadine), Hismanal (astemizole), Propulsid (cisapride) within 1 month prior to dosing MK-0974 or placebo and throughout the study period; participant has received an investigational medication within 4 weeks prior to the prestudy (screening) visit.
* Participant has a history of multiple and/or severe allergies, or has had an anaphylactic reaction or intolerability to prescription or non-prescription drugs or food.
* There is any concern by the investigator regarding the safe participation of a participant in the study, or for any other reason the investigator considers the participant inappropriate to participate in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-02-12 (Actual); Primary Completion 2009-02-28 (Actual); Study Completion 2009-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Chaitman BR, Ho AP, Behm MO, Rowe JF, Palcza JS, Laethem T, Heirman I, Panebianco DL, Kobalava Z, Martsevich SY, Free AL, Bittar N, Chrysant SG, Ho TW, Chodakewitz JA, Murphy MG, Blanchard RL. A randomized, placebo-controlled study of the effects of telcagepant on exercise time in patients with stable angina. Clin Pharmacol Ther. 2012 Mar;91(3):459-66. doi: 10.1038/clpt.2011.246. Epub 2012 Jan 25. PMID 22278333
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0974-014&kw=0974-014&tab=access

RESULTS

PARTICIPANT FLOW:
Groups:
- Telcagepant Then Placebo: Participants receive single oral dose of 600 mg (two 300 mg capsules or two bioequivalent 280 mg tablets) or 900 mg telcagepant (three 300 mg capsules) in Period 1 and single oral dose of two capsules or tablets of placebo for telcagepant (or three capsules of placebo for telcagepant) in Period 2 of the crossover. Each treatment period is separated by a washout of 96-240 hours.
- Placebo Then Telcagepant: Participants receive single oral dose of two capsules or tablets of placebo for telcagepant (or three capsules of placebo for telcagepant) in Period 1 and a single oral dose of 600 mg (two 300 mg capsules or two bioequivalent 280 mg tablets) or 900 mg telcagepant (three 300 mg capsules) in Period 2 of the crossover. Each treatment period is separated by a washout of 96-240 hours.
Period: Period 1
Arm/Group | Telcagepant Then Placebo | Placebo Then Telcagepant
Started | 31 | 33
Completed | 30 | 32
Not Completed | 1 | 1
Period: Washout Period
Arm/Group | Telcagepant Then Placebo | Placebo Then Telcagepant
Started | 30 | 32
Completed | 29 | 31
Not Completed | 1 | 1
Period: Period 2
Arm/Group | Telcagepant Then Placebo | Placebo Then Telcagepant
Started | 29 | 31
Completed | 28 | 31
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of study drug.
Groups:
- All Enrolled Participants: All enrolled participants who recieved at least one dose of either telcagepant or placebo.
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 64
Age, Continuous [Mean (Full Range); unit: years] | 63.5 (10.38) [38 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 55

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Adverse Events (AEs)
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the product, was also an AE. A clinical AE was an AE reported as a result of a clinical examination or reported by the participant.
Time Frame: Up to 10 days post dose in Period 1 and up to 14 days post dose in Period 2
Population: Safety Population which consisted of all enrolled participants who actually received assigned study drug in a particular period . Adverse events are reported by dose taken in a given treatment period and not by randomly assigned treatment sequence.
Measure: Number; unit: Participants
Groups:
- Telcagepant (600 mg): Participants who received a single oral dose of 600 mg telcagepant capsules (or 560 mg of bioequivalent tablets) in Period 1 or 2 of crossover
- Telcagepant (900 mg): Participants who received a single oral dose of 900 mg telcagepant in Period 1 or 2 of crossover
- Placebo: Participants who received a single oral dose of placebo in Period 1 or 2 of crossover
Arm/Group | Telcagepant (600 mg) | Telcagepant (900 mg) | Placebo
Number analyzed (Participants) | 46 | 16 | 62
Participants | 7 | 1 | 5

2. Primary Outcome: Number of Participants With Laboratory Adverse Events
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the product, was also an AE. A laboratory AE was an AE reported as a result of a laboratory assessment or test.
Time Frame: Up to 10 days post dose in Period 1 and up to 14 days post dose in Period 2
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Telcagepant (600 mg) | Telcagepant (900 mg) | Placebo
Number analyzed (Participants) | 46 | 16 | 62
Participants | 0 | 0 | 0

3. Primary Outcome: Total Exercise Duration on the Treadmill Test
Description: Bruce (and Modified Bruce) Protocol was used to assess the exercise duration on a treadmill. This protocol consists of a standardized gradual incremental increase in external workload every 3 minutes while the participant's electrocardiogram (ECG), symptoms, and arm blood pressure were continuously monitored. Regardless of whether the participant believed he or she could continue, the test was discontinued upon evidence of chest discomfort, severe shortness of breath, dizziness, fatigue, ST-segment depression of greater than 2 mm, a fall in systolic blood pressure exceeding 10 mmHg, or the development of a ventricular tachyarrhythmia
Time Frame: 2.5 to approximately 2.75 hours post dose of each treatment period
Population: Enrolled participants with evaluable treadmill exercise duration data available. Data from the 600 and 900 mg telcagepant treatments were grouped for comparsion to placebo.
Measure: Least Squares Mean (95% Confidence Interval); unit: Seconds
Groups:
- Telcagepant: Participants who received a single oral dose of 600 mg (or bioequivalent 560 mg tablets) or 900 mg telcagepant in Period 1 or 2 of crossover
- Placebo: Participants who received single oral dose of placebo in Period 1 or 2 of crossover
Arm/Group | Telcagepant | Placebo
Number analyzed (Participants) | 60 | 58
Seconds | 405.38 [375.91 to 434.85] | 412.28 [382.72 to 441.85]
Statistical Analysis 1: Comparison: Telcagepant vs Placebo; Telcagepant minus Placebo Treatment Difference; Test type: Superiority or Other; mixed effects model; mixed effects model with MK-0974 pooled over doses; Difference in Least Squares Means = -6.90, 90% CI 2-sided [-17.66 to 3.86]

4. Secondary Outcome: ST Segment Depression at Peak Exercise
Description: Bruce (and Modified Bruce) Protocol was used to assess the exercise duration on a treadmill. This protocol consists of a standardized gradual incremental increase in external workload every 3 minutes while the participant's ECG, symptoms, and arm blood pressure were continuously monitored. The time of peak exercise was considered the time at which the participant reached at least one of the criteria for stopping the treadmill test (evidence of chest discomfort, severe shortness of breath, dizziness, fatigue, ST-segment depression of greater than 2 mm, a fall in systolic blood pressure exceeding 10 mmHg, or the development of a ventricular tachyarrhythmia). The ECG for that timepoint (time of peak exercise) was evaluated and the amount of ST segment depression was determined.
Time Frame: 2.5 to approximately 2.75 hours post dose of each treatment period
Population: Enrolled participants with evaluable data for assessment of ST segment depression at peak exercise available. Data from the 600 and 900 mg telcagepant treatments were grouped for comparsion to placebo.
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | Telcagepant | Placebo
Number analyzed (Participants) | 57 | 55
mm | -1.91 [-2.13 to -1.70] | -1.86 [-2.08 to -1.64]
Statistical Analysis 1: Comparison: Telcagepant vs Placebo; Telcagepant minus Placebo Treatment Difference; Test type: Superiority or Other; mixed effects model; mixed effects model with MK-0974 pooled over doses; Difference in Least squares meand = -0.056, 90% CI 2-sided [-0.19 to 0.076]

5. Secondary Outcome: Time to 1 mm ST Segment Depression
Description: Bruce (and Modified Bruce) Protocol was used to assess the exercise duration on a treadmill. This protocol consists of a standardized gradual incremental increase in external workload every 3 minutes while the participant's ECG, symptoms, and arm blood pressure were continuously monitored. The ECG was reviewed and the time to the first ST segment depression of 1 mm was recorded.
Time Frame: 2.5 to approximately 2.75 hours post dose of each treatment period
Population: Enrolled participants with evaluable data for assessment of time to 1 mm ST segment depression available. Data from the 600 and 900 mg telcagepant treatments were grouped for comparsion to placebo.
Measure: Least Squares Mean (95% Confidence Interval); unit: seconds
Arm/Group | Telcagepant | Placebo
Number analyzed (Participants) | 57 | 56
seconds | 363.53 [330.78 to 396.27] | 370.67 [337.85 to 403.49]
Statistical Analysis 1: Comparison: Telcagepant vs Placebo; Telcagepant minus Placebo Treatment Difference; Test type: Superiority or Other; mixed effects model; mixed effects model with MK-0974 pooled over doses; Difference in Least Squares Means = -7.14, 90% CI 2-sided [-22.03 to 7.74]

ADVERSE EVENTS:
Time Frame: Up to 10 days post dose in Period 1 and up to 14 days post dose in Period 2
Description: AEs are reported by dose taken in a given treatment period and not by randomly assigned treatment sequence.
Arm/Group | Telcagepant (600 mg) | Telcagepant (900 mg) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/16 | 0/62
Other Adverse Events (participants affected / at risk) | 0/46 | 1/16 | 0/62
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Telcagepant (600 mg) (N=46) | Telcagepant (900 mg) (N=16) | Placebo (N=62)
Feeling Jittery (General disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications derived from this study should include input from the investigator(s), and SPONSOR personnel. The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication guidelines.